CLINICAL TRIAL: NCT04720820
Title: A Pragmatic Multicenter Randomized Controlled Study on Early Supported Discharge: KOrean Model of Post-Acute Comprehensive rehabiliTation(KOMPACT)
Brief Title: Efficacy and Safety of Early Supported Discharge for Post-Acute Stroke Patients in Korea
Acronym: KOMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Chungnam National University Hospital (Other); Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Nam-Jong Paik, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-2012-654-308
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2023-11

CONDITIONS: Stroke
Keywords: Early Supported Discharge; Acute stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The trial consists of two arms; An Early Supported Discharge group and Conventional Rehabilitation group
Who Masked: Outcomes Assessor
Masking Description: The assessors are blinded to the patients' group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Supported Discharge (ESD) Group (Experimental): Patients in the ESD group will be discharged to home as soon as the acute medical treatment is finished. The patients will follow a pre-planned ESD program which consists of home-based rehabilitation (at least 30 minutes of physical therapy and 30 minutes of occupational therapy per week) offered by therapists. The ESD team will also provide social/medical services as needed. The ESD program will be provided till 1 months after discharge point.
  Interventions: Other: Early Supported discharge with home based Rehabilitation
- Conventional Rehabilitation (CR) Group (Active Comparator): The patients in CR group will be provided with inpatient rehabilitation after the acute medical treatment is finished. The length of inpatient rehabilitation may depend on the hospital's current program. Patients will be provided with outpatient based rehabilitation program if needed after discharge.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Other: Early Supported discharge with home based Rehabilitation — Treatment by Physiotherapist and occupational therapist at least 30 minutes each, per week provided at home.
  Arms: Early Supported Discharge (ESD) Group
Other: Conventional rehabilitation — Treatment will be provided according to current hospital's stroke rehabilitation program.
  Arms: Conventional Rehabilitation (CR) Group

SUMMARY:
The study aims to examine the effect of early supported discharge (ESD) service on the functional outcomes and quality of life of acute stroke patients with mild to moderate disability in Korea.

The study is a double-armed prospective multi-centered, assessor-blinded randomized controlled trial comparing the effect of ESD program with conventional rehabilitation program.

DETAILED DESCRIPTION:
Early Supported Discharge (ESD) is a form of medical service applicable to acute stroke patients with mild to moderate disabilities. ESD service was developed to facilitate patient to their daily livings at home, reduce the length of stay in the hospital with possibly better or equivalent outcomes for patients and caregivers.

ESD service has been proven to be non-inferior in the functional and quality of life measures as well as cost-effective, compared to the conventional rehabilitation service in many countries, however the effectiveness of ESD service may differ among countries and medical, economical circumstances. This study aims to examine the effect of ESD service on the acute stroke patients with mild to moderate disabilities in Korea and demonstrate its feasibility as an alternative medical service option to those patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is over 20 years old
* Patient who had acute stroke and admitted to hospital (excludes TIA)
* Patient who will be discharged to home within 30 days after onset
* Patient who has indwelling caregiver and is able to support in ESD program
* Patient who's initial mRS is 1-3
* Patient who's initial FAC is 3 or above
* Patient who's initial K-NIHSS consciousness scores (1a,1b,1c) are all 0

Exclusion Criteria:

* Patient who had Transient Ischemic Attack
* Patient who is medically unstable requiring intense treatment
* Patient who has indwelling urinary catheter
* Patient who is unable to intake food by mouth
* Patient who is initial MMSE is below 15
* Patient who has uncontrolled pain
* Patient who has psychobehavioral problems

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
changes in Korean modified Barthel Index (K-MBI) | Baseline, 1 month after discharge, 3 months after onset, changes from baseline
  K-MBI is an ordinal scale used to measure performance in activities of daily living(ADL). score ranges from 0 to 100, higher score meaning better ADL function.

SECONDARY OUTCOMES:
modified Rankin Scale (mRS) | Baseline, 1 month after discharge, 3 months after onset
  mRS is a scale used for measuring the degree of disability or dependence in the daily activities of people with stroke. Scale ranges from 0-6, with 0 meaning no symptoms and 6 meaning dead.
Korean Instrumental Activities of Daily Living (K-IADL) | 1 month after discharge, 3 months after onset
  K-IADL assesses a person's ability to perform tasks such as using a telephone, doing laundry, and handling finances. The scale ranges from 0 to 100, higher score meaning better IADL function.
Korean Reintegration to Normal Life Index (K-RNLI) | 1 month after discharge, 3 months after onset
  K-RNLI assesses the degree of individuals who have experienced stroke achieve reintegration into normal social activities. The scale ranges from 0-100 with higher score meaning better reintegration to normal life.
Patient Health Questionnaire-9 (PHQ-9) | Baseline, 1 month after discharge, 3 months after onset
  PHQ-9 is a instrument for screening, diagnosing and measuring the severity of depression. The scale ranges from 0-27 with higher score indicating severer depression.
Korean Stroke Impact Scale ver 3.0 (K-SIS) | 1 month after discharge, 3 months after onset
  K-SIS evaluates disability and health-related quality of life after stroke. It consists of 8 domains each score ranges from 0-100 with higher score meaning better quality of life.
European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) | Baseline, 1 month after discharge, 3 months after onset
  EQ-5D-5L evaluates the quality of life. The scale ranges from -0.066 to 0.904, lower value means worse quality of life.
Fall Experience | 1 month after discharge, 3 months after onset
  Number of patients who experience fall within the period.
Mortality rate | 1 month after discharge, 2 month after discharge(if needed), 3 months after onset
  Number of patients who died within the period.
Readmission rate | 1 month after discharge, 2 month after discharge(if needed), 3 months after onset
  Number of patients who were readmitted to the hospital within the period.
Length of hospital stay | 3 months after onset
  Number of days admitted to hospital for stroke treatment and post-stroke rehabilitation.
Korean Zarit Burden Interview-22 (K-ZBI 22) | 1 month after discharge, 3 months after onset
  K-ZBI 22 assesses caregiver perceptions of burden in health, personal, social or financial domains. The scale ranges from 0-88 with higher score indicating higher burden.
Direct costs related to rehabilitation | 1 month after discharge, 2 month after discharge(if needed), 3 months after onset
  Direct costs includes expenses for medical and rehabilitation services. It consists for inpatient cost, outpatient cost, home based rehabilitation cost.
Indirect costs related to rehabilitation | 1 month after discharge, 2 month after discharge(if needed), 3 months after onset
  Indirect costs means expenses needed for treatment and rehabilitation of the patients other tahn medical and rehabilitation services. Indirect costs include transportation expense and caregiver expense and productivity loss

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam-si, Korea, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chang WK, Jung YS, Choi JS, Kim WS, Sohn MK, Jee S, Shin YI, Ko SH, Ock M, Kim HJ, Paik NJ. Pragmatic multicenter randomized controlled study on early supported discharge after stroke in Korea: the KOMPACT study. Ann Phys Rehabil Med. 2025 Nov;68(8):102025. doi: 10.1016/j.rehab.2025.102025. Epub 2025 Sep 18. PMID 40972310
- [Derived] Chang WK, Kim WS, Sohn MK, Jee S, Shin YI, Ko SH, Ock M, Kim HJ, Paik NJ. Korean Model for Post-acute Comprehensive rehabilitation (KOMPACT): The Study Protocol for a Pragmatic Multicenter Randomized Controlled Study on Early Supported Discharge. Front Neurol. 2021 Sep 8;12:710640. doi: 10.3389/fneur.2021.710640. eCollection 2021. PMID 34566853